CLINICAL TRIAL: NCT00950690
Title: Observational Study Assessing The Efficacy And Tolerability Of Xalatan™ In Patients With Open Angle Glaucoma And /Or Ocular Hypertension.
Brief Title: Efficacy and Tolerability of Xalatan in Patients
Acronym: A6111128
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6111128; A6111128
Record Dates: First submitted 2009-03-31; First posted 2009-08-03 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2011-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: observational safety study
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Drug - Xalatan 0.005% eye drops
  Interventions: Drug: Xalatan 0.005% eye drops

INTERVENTIONS:
Drug: Xalatan 0.005% eye drops — ophthalmic solution dosed once daily for 3 months
  Other Names: latanoprost

SUMMARY:
Efficacy data was not collected or analyzed. This study did assess safety and tolerability of Xalatan.

DETAILED DESCRIPTION:
* Efficacy data not collected or analyzed
* Safety and tolerability of Xalatan assessed NA

ELIGIBILITY:
Inclusion Criteria:

* Patient with ocular hypertension at least 22mg Hg
* Patient must be over 18 years old

Exclusion Criteria:

* None listed in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with glauocma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1289 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Alexandria, Egypt
- Pfizer Investigational Site, Jeddah, Saudi Arabia
- Pfizer Investigational Site, Umm Al Quwain City, United Arab Emirates

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111128&StudyName=efficacy%20and%20tolerability%20of%20Xalatan%20in%20patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigative sites
Groups:
- Xalatan: 0.005% ophthalmic solution dosed once daily for 3 months
Period: Overall Study
Arm/Group | Xalatan
Started | 1349
Completed | 1105
Not Completed | 244
Not completed — Death | 4
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 22
Not completed — Lost to Follow-up | 40
Not completed — Other | 163

BASELINE CHARACTERISTICS:
Arm/Group | Xalatan
Number analyzed (Participants) | 1349
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.0)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 723
  Female | 584
  Unspecified | 42

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intraocular pressure was measured at each visit
Time Frame: Screening, 10 days, 4 weeks and 12 weeks after beginning treatment
Population: Data collection process did not permit clear identification of IOP & visual field data in non-monitored study. Efficacy data not sufficiently interpretable for statistical summaries.
Arm/Group | Xalatan
Number analyzed (Participants) | 0

2. Primary Outcome: Humphrey Perimetry Visual Field
Description: Analysis of visual field deficits for abnormalities.
Time Frame: Visits 1 and 4
Population: as for outcome 1
Arm/Group | Xalatan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Xalatan
Serious Adverse Events (participants affected / at risk) | 5
Other Adverse Events (participants affected / at risk) | 101
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Xalatan
Iridocyclitis (Eye disorders) | 1/1349
Retinal detachment (Eye disorders) | 1/1349
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/1349
Hypoglycaemic coma (Nervous system disorders) | 1/1349
Erythema (Skin and subcutaneous tissue disorders) | 1/1349
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Xalatan
Palpitations (Cardiac disorders) | 1/1349
Ear Pain (Ear and labyrinth disorders) | 1/1349
Conjunctival follicles (Eye disorders) | 1/1349
Conjunctival hyperaemia (Eye disorders) | 7/1349
Conjunctivitis (Eye disorders) | 2/1349
Corneal erosion (Eye disorders) | 2/1349
Dry eye (Eye disorders) | 4/1349
Eye disorder (Eye disorders) | 4/1349
Eye irritation (Eye disorders) | 1/1349
Eye pain (Eye disorders) | 1/1349
Glaucoma (Eye disorders) | 1/1349
Ocular hyperaemia (Eye disorders) | 7/1349
Uveitis (Eye disorders) | 1/1349
Condition aggravated (General disorders) | 1/1349
Drug effect decreased (General disorders) | 1/1349
Drug ineffective (General disorders) | 1/1349
Ill-defined disorder (General disorders) | 22/1349
Pain (General disorders) | 1/1349
Human ehrlichiosis (Infections and infestations) | 1/1349
Intraocular pressure increased (Investigations) | 1/1349
Back pain (Musculoskeletal and connective tissue disorders) | 1/1349
Burning sensation (Nervous system disorders) | 1/1349
Headache (Nervous system disorders) | 1/1349
Asthma (Respiratory, thoracic and mediastinal disorders) | 2/1349
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/1349
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1/1349
Erythema (Skin and subcutaneous tissue disorders) | 9/1349
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3/1349
Hyperaemia (Vascular disorders) | 19/1349
Hypertension (Vascular disorders) | 1/1349
Vertigo (Ear and labyrinth disorders) | 1/1349

LIMITATIONS AND CAVEATS:
Efficacy data were not summarized or analyzed because data collection did not permit clear identification of IOP & visual field data in this non-monitored observational study. Consequently, data were not sufficiently interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.